CLINICAL TRIAL: NCT01948648
Title: Effects of Fish Oil, Colesevelam and Combination Therapy on Sterol Metabolism in Sitosterolemia
Brief Title: Effects of Fish Oil and Colesevelam (STAIR7007)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: B2013:075
Record Dates: First submitted 2013-09-06; First posted 2013-09-23 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2019-12

CONDITIONS: Sitosterolemia
Keywords: plant sterols; cholesterol; colesevelam; phytosterolemia; fish oil
MeSH Terms: conditions — Sitosterolemia | interventions — Colesevelam Hydrochloride; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colesevelam (Active Comparator): 3.75g/day for 6 weeks
  Interventions: Drug: Colesevelam
- Fish Oil (Active Comparator): 1g/day for 6 weeks
  Interventions: Dietary Supplement: Fish Oil
- Combination of Fish Oil and Colesevelam (Active Comparator): 3.75g/day of colesevelam and 1g/day of fish oil for 6 weeks
  Interventions: Drug: Combination of fish oil and colesevelam

INTERVENTIONS:
Drug: Colesevelam — Drug is in powder form, each packet contains 3.75g of colesevelam hydrochloride. Participant will mixed it with water and have 1 packet per day during the treatment session.
  Other Names: Lodalis
  Arms: Colesevelam
Dietary Supplement: Fish Oil — In softgel form, contains 660mg EPA and 330mg DHA. Participant consume 1 softgel per day during treatment session.
  Other Names: Omega-3
  Arms: Fish Oil
Drug: Combination of fish oil and colesevelam — combination of both colesevelam and fish oil. Participant will consume 1 packet and 1 softgel per day during treatment session.
  Other Names: Omega-3 and Lodalis
  Arms: Combination of Fish Oil and Colesevelam

SUMMARY:
If treatment of colesevelam, fish oil in conjunction with ezetimibe, will lead to further reduction in plasma plant sterol levels in sitosterolemia patients. We hypothesize that treatments with fish oil, colesevelam and ezetimibe will maximize decrease in plasma concentrations of sitosterol and other plant sterols in sitosterolemia patients.

DETAILED DESCRIPTION:
Ezitimibe significantly lowers plant sterol levels in the blood of patients with sitosterolemia. However, plant sterol levels remain substantially elevated compared to those in healthy individuals. Thus, combination therapy needs to be considered. Agents that provide cardiovascular benefits such as colesevelam, a second-generation bile acid sequestrant, and fish oil are potential candidates to help further reduce sterol levels, but have yet to be evaluated in sitosterolemia patients.

The purpose of this study is to dtermine the effects of colesevelam, fish oil and combination therapy (fish oil + colesevelam) on plant sterols, cholesterol and cardiovascular risk factors in sitosterolemia patients treated with ezetimibe. The results of this study will enhance knowledge on the pathogenesis of sitosterolemia and the mechanisim of actions of colesevelam and fish oil as adjunct therapies to ezitimibe in patients with the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of homozygous sitosterolemia as established by genotyping and/or clinical parameters
2. Receiving ezetimibe treatment
3. Over 8 years of age (no maximum)
4. Concomitant illnesses or conditions

Exclusion Criteria:

1. Pregnancy
2. Intellectual disability
3. Bowel or biliary obstruction
4. Known hypersensitivity to colesevelam or any ingredients of colesevelam

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Plasma plant sterol level | 32 weeks
  plasma plant sterol assessment using Gas Chromatography(GC)

SECONDARY OUTCOMES:
Fatty acid | 32 weeks
  use of gas chromatography technique to measure fish oil intervention
endothelial functions | 32 weeks
  use of EndoPAT 2000 system to assess endothelial function

CONTACTS AND LOCATIONS:
Locations (1):
- Richardson Center for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada